CLINICAL TRIAL: NCT06886568
Title: Ultrasound Guided Ganglion Impar Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Tuba Tanyel Saraçoğlu, MD, Head of Algology Department, Başakşehir Çam & Sakura City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022.03.98
Record Dates: First submitted 2025-03-03; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Coccydynia; Chronic Pain
Keywords: Coccydynia; pain; ultrasound guided injection; ganglion impar
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Injection Group (Experimental): Ganglion impar block will be applied under ultrasound guidance
  Interventions: Procedure: Ultrasound-guided ganglion impar block

INTERVENTIONS:
Procedure: Ultrasound-guided ganglion impar block — The procedure will be performed under sterile conditions and continuous monitoring. Using an ultrasound device with a 10-12 MHz linear probe, a 22G spinal needle will be advanced into the sacrococcygeal joint space using the out-of-plane technique. After confirming loss of resistance with a syringe containing normal saline as the needle exits the capsule anterior to the joint, approximately 1 mL of contrast medium will be injected. Anteroposterior (AP) and lateral fluoroscopic images will be obtained to verify the spread of the contrast agent. Once adequate contrast distribution is confirmed anterior to the coccyx on the lateral view, a mixture of dexamethasone and bupivacaine will be injected to complete the block. Procedures that cannot be completed or successfully visualized under ultrasound guidance will be finalized under fluoroscopic guidance.

SUMMARY:
The aim of this study is to evaluate feasibility, reliability and short term effectiveness of ganglion impar block with ultrasound in patients with chronic coccygodinia.

DETAILED DESCRIPTION:
Ganglion impar blocks have long been used for coccydynia, either with a landmark-based technique or fluoroscopic guidance. With the growing use of ultrasound, ultrasound-guided ganglion impar block has become a viable alternative.

Despite its frequent use in clinical practice, ultrasound has limitations in visualizing structures behind the bone, while fluoroscopy remains the gold standard. Further research is needed to evaluate its feasibility, safety, and efficacy.

This study primarily aims to assess the feasibility and safety of ultrasound-guided ganglion impar block in coccydynia. Additionally, it will examine its short-term (1-month) efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years.
* Coccydynia persisting for at least three months.
* Being scheduled for a ganglion impar block in the pain medicine outpatient clinic.
* Having inadequate response to medical and conservative treatments.
* Aggreeing to undergo the interventional procedure and participate in the study.

Exclusion Criteria:

* Local infection at the injection site.
* Bleeding disorders or diseases and drugs that may cause bleeding diatesis (e.g. renal failure, liver failure, anticoagulant treatments)
* History of allergic reaction to the medications to be used.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Injection accuracy | Post-procedure 1st hour
  In all patients, the sacrococcygeal or transcoccygeal space will be identified under ultrasound guidance. A 22-gauge spinal needle will be advanced into the joint space under ultrasound visualization. Using a saline-filled syringe, the loss-of-resistance technique will be employed to confirm passage through the joint space and entry into the retroperitoneal space. Subsequently, a lateral fluoroscopic image will be obtained, and contrast medium will be injected to verify needle placement. If appropriate contrast dispersion is observed along the midline, the procedure will be considered successful, and the medication will be administered. If contrast distribution is inadequate (e.g. vascular spread, non-midline spread), the procedure will be discontinued under ultrasound guidance and resumed under fluoroscopic guidance.

SECONDARY OUTCOMES:
Visual Analogue Scale | Baseline, 1st hour, 1st week, 1st month
  Pain intensity will be assessed using the Visual Analogue Scale (VAS), a 10-point scale where 1 indicates no pain and 10 represents the worst pain.
Pain-free sitting duration | Baseline, 1st hour, 1st week, 1st month
  Pain-free sitting duration (minutes) will be recorded.
The number of attempts | Post-procedure 1st hour
  The number of attempts will be recorded.
Technical difficulty of injection | Post-procedure 1st hour
  The technical difficulty of the injection will be assessed using a 10-item scale, where 1 indicates no difficulty and 10 represents the highest level of difficulty
Complications | Baseline, 1st hour, 1st week, 1st month
  All complications following the injection will be recorded, including infections, bleeding, hematoma, allergic reactions, steroid-related complications, transient hypoesthesia, and weakness, among others.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Karali-Bingul, MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Başakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li SQ, Jiang L, Cui LG, Jia DL. Clinical efficacy of ultrasound-guided pulsed radiofrequency combined with ganglion impar block for treatment of perineal pain. World J Clin Cases. 2021 Mar 26;9(9):2153-2159. doi: 10.12998/wjcc.v9.i9.2153. PMID 33850934
- [Background] Ghai A, Jangra P, Wadhera S, Kad N, Karwasra RK, Sahu A, Jaiswal R. A prospective study to evaluate the efficacy of ultrasound-guided ganglion impar block in patients with chronic perineal pain. Saudi J Anaesth. 2019 Apr-Jun;13(2):126-130. doi: 10.4103/sja.SJA_667_18. PMID 31007658
- [Background] Lin CS, Cheng JK, Hsu YW, Chen CC, Lao HC, Huang CJ, Cheng PH, Narouze S. Ultrasound-guided ganglion impar block: a technical report. Pain Med. 2010 Mar;11(3):390-4. doi: 10.1111/j.1526-4637.2010.00797.x. PMID 20447308